CLINICAL TRIAL: NCT07300254
Title: Treponemal Shedding, Load, and Viability, in Women and Men-who-have-sex-with-women Only With Early Infectious Syphilis: Implications for Transmission
Brief Title: Treponemal Shedding, Load, and Viability, in Women and Men-who-have-sex-with-women-only With Early Infectious Syphilis: Implications for Transmission
Acronym: SOS Global
Status: Recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: Melbourne Sexual Health Centre (Unknown); The Alfred (Other)
Responsible Party: Sponsor
Other Study IDs: MUCTC-24018
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Syphilis
Keywords: syphilis; sexual health; syphilis transmission; asymptomatic shedding
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — genital swabs, urine sample, blood sample, anal swab, oral swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cis-women with suspected or confirmed primary syphilis infection: Cis-women with suspected or confirmed primary syphilis infection
  Interventions: Other: No Intervention: Observational Cohort
- Cis-women with suspected or confirmed secondary syphilis infection: Cis-women with suspected or confirmed secondary syphilis infection
  Interventions: Other: No Intervention: Observational Cohort
- Cis-women with confirmed early-latent syphilis infection: Cis-women with confirmed early-latent syphilis infection
  Interventions: Other: No Intervention: Observational Cohort
- Men-who-have-sex-with-women-only with suspected or confirmed primary syphilis infection: Men-who-have-sex-with-women-only with suspected or confirmed primary syphilis infection
  Interventions: Other: No Intervention: Observational Cohort
- Men-who-have-sex-with-women-only with suspected or confirmed secondary syphilis infection: Men-who-have-sex-with-women-only with suspected or confirmed secondary syphilis infection
  Interventions: Other: No Intervention: Observational Cohort
- Men-who-have-sex-with-women-only with confirmed early-latent syphilis infection: Men-who-have-sex-with-women-only with confirmed early-latent syphilis infection
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention: Observational study

SUMMARY:
How syphilis is transmitted between sexual partners is unclear. Asymptomatic detection i.e. detection of syphilis bacteria (Tp) from anatomical sites without lesions, in patients with syphilis infection, suggests that asymptomatic transmission from these sites may play a role. However, no existing studies have established whether the syphilis bacteria (Tp) detected was viable. This means it is not known if the bacteria at this anatomical site is alive and therefore able to transmit the infection. Further, studies have focused mostly on men who have sex with men, resulting in a lack of evidence regarding anal shedding in men-who-have-sex-with-women only and women (regardless of sexual behaviour), and no data on asymptomatic vaginal shedding in women. This study will explore:

1. Patterns of Tp detection in women and men-who-have-sex-with-women only.
2. Whether detected Tp from each asymptomatic anatomical sites is viable
3. Duration of Tp detection and viability (alive and transmissible bacteria). Patients presenting to a participating sexual health service (overseas only) for management of suspected/confirmed early infectious syphilis will be eligible. During the routine clinical examination, participants will have additional oral and anal swabs, urine, vaginal swab (where relevant), penile skin swab (where relevant) and blood sample collected, in addition to the routine samples taken from the same sites and routine serology collected when syphilis is diagnosed.

ELIGIBILITY:
Inclusion Criteria:

- 1. Any cis-woman, cis-MSW, or nonbinary individuals with a penis who have sex with women only, (who meet all other study criteria) 2. Aged ≥18 years of age, 3. At least one sexual partner in the last 12 months 4. One of either:

a. Untreated clinically suspected primary or secondary syphilis. i. Must have rash or lesion(s) clinically suggestive of early infectious syphilis infection.

ii. May have positive PCR result, positive Dark-ground Microscopy result, positive syphilis serology or positive point-of-care syphilis test, but these are not necessary at the time of enrolment.

b. Untreated early latent (no clinical signs indicative of primary or secondary syphilis) syphilis with positive syphilis serology or positive point-of-care test, and one or more of the following(11): i. A documented syphilis seroconversion within the prior 12 months. ii. A sustained (longer than 2 weeks) fourfold or greater increase in the titre in the prior 12 months in a person previously treated for syphilis.

iii. Unequivocal symptoms of primary or secondary syphilis within the prior 12 months.

iv. Contact in the prior 12 months with a sex partner who had untreated primary, secondary, or early latent syphilis.

v. Documented reactive nontreponemal and treponemal tests, and the only possible exposure occurred during the previous 12 months vi. RPR/VDRL titre >= 1:64 5. Be willing and able to complete study procedures, including physical examination 6. Receiving syphilis treatment on the day of recruitment 7. Have sufficient language proficiency to understand the requirements of the study 8. Provide informed consent as per individual site's local ethics requirements

Exclusion Criteria:

1. Men, transwomen, or other people, with a penis, who have had any sexual contact, including kissing, oral sex or anal sex, with men (or any other individual with a penis) in the previous one year.
2. Individuals who have received antibiotic treatment within 1 month prior to enrolment, with the EXCEPTION of metronidazole.
3. Diagnosis of late latent syphilis (>1 year) or latent syphilis of unknown duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Unfortunately we are unable to accept people who identify as transgender
Study Population: Women and Men-Who-Have-Sex-With-Women-Only with early infectious syphilis
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Biological Samples Testing Positive for Treponema pallidum DNA by PCR | Samples are taken at time of consent - single visit study
  This outcome measures the presence of Treponema pallidum (Tp) DNA in collected biological samples-including lesion swabs, blood, urine, saliva, and oral/anal/genital swabs-using a validated T. pallidum polymerase chain reaction (Tp PCR) assay.
  Data will be reported as the number and proportion of samples that test positive, stratified by:
  * sample type,
  * clinical stage of syphilis,
  * anatomical site (where applicable),
  * and participant characteristics relevant to the SOS Global protocol. No scale is used; this is a binary laboratory outcome (PCR positive / PCR negative).

SECONDARY OUTCOMES:
Load of Treponema pallidum DNA in Positive Biological Samples by In-house Quantitative PCR (qPCR) assay | Samples are taken at time of consent - single visit study
  This outcome measures the load (copies/mL) of Treponema pallidum (Tp) DNA in collected biological samples-including lesion swabs, blood, urine, saliva, and oral/anal/genital swabs-using an in-house validated quantitative T. pallidum polymerase chain reaction (Tp qPCR) assay.
  Data will be reported as a comparison in load between anatomical sites and by clinical stage of syphilis.
Number of Treponema pallidum-Positive Samples Demonstrating Viable Organisms via Novel In-house Viability Assay | Samples are collected at time of consent - single study visit
  This outcome measures the viability of detected Treponema pallidum in PCR-positive biological samples. Viability is assessed using a novel in-house viability assay.
  Results will be summarised as the number and proportion of Tp PCR-positive samples that contain viable organisms, stratified by sample type and clinical/epidemiological variables specified in the SOS Global protocol.
  This outcome focuses on confirming whether Tp organisms in collected specimens are capable of establishing infection, rather than merely detecting genetic material. The viability assessment does not result in a continuous scale; it is a binary laboratory outcome (viable / non-viable).

CONTACTS AND LOCATIONS:
Overall Officials: Janet Towns, Principal Investigator — Monash University
Locations (8):
- Monash University, Melbourne, Victoria, Australia
- China (2):
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
- Foundation for Professional Development, Pretoria, South Africa
- United Kingdom (4):
  - Burrell Street Clinic, Guy's and St Thomas', London
  - Jefferiss Clinic St Mary's Hospital, Imperial College London, London
  - Mortimer Market Centre, London
  - London School of Hygiene & Tropical Medicine, London

IPD SHARING:
Plan to Share IPD: Undecided
Request for data sharing will be considered on a case by case basis